CLINICAL TRIAL: NCT01860937
Title: A Phase I Trial of T-Lymphocytes Genetically Targeted to the B-Cell Specific Antigen CD19 in Pediatric and Young Adult Patients With Relapsed B-Cell Acute Lymphoblastic Leukemia
Brief Title: T-Lymphocytes Genetically Targeted to the B-Cell Specific Antigen CD19 in Pediatric and Young Adult Patients With Relapsed B-Cell Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13-052
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Relapsed B-Cell Acute Lymphoblastic Leukemia
Keywords: T cell Immunotherapy; CD19 Targeted Therapy; Chimeric Antigen Receptor (CAR) Modified T cells; Conditioning Chemotherapy; 13-052
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Leukapheresis

ARMS (2):
- Cohort 1 (MRD) (Experimental): Patients with no morphologic evidence of disease at the time of T cell infusion, (<5% blasts in the bone marrow) as assessed by morphology or flow cytometry. Participating site PI to determine cohort stratification in the event of morphology/flow cytometry blast count discrepancy. Cohort 1 patients will receive conditioning chemotherapy followed by 1x10^6 19-28z+ T cells/kg over 1 to 2 days. During formulation of End of Production (EOP) T cells, under or over estimation of CAR modified T-cells may occur. Patients may receive an altered fractionation of the total doses (e.g. ½ on Day 0 and ½ on Day +1) or up to 35% over total cell dose with approval by the participating site PI. In both cohorts, patients will be allowed to receive a 2nd treatment of 19-28z+ T cells if they benefited from the first infusion and did not experience any non-hematologic grade 4 toxicities.
  Interventions: Procedure: leukapheresis or collection of PBMCs; Drug: cyclophosphamide based chemotherapy regimens; Biological: modified T cells
- Cohort 2 (Morphologic Disease) (Experimental): Pts with morphologic evidence of disease at the time of T cell infusion, (≥5% blasts in the bone marrow) as assessed by morphology or flow cytometry. Participating site PI to determine cohort stratification in the event of morphology/flow cytometry blast count discrepancy. Pts with increased blasts (5-10% blasts) that are immunophenotypically consistent with recovering marrow from prior re-induction chemo may be treated under Cohort 1 with approval of the participating site PI. Cohort 2 pts will get conditioning chemo followed by 1x10^6 19-28z+ T cells/kg over 1 to 2 days. During formulation of EOP T cells, under or over estimation of CAR modified T-cells may occur. Pts may get up to 35% over total cell dose with approval by the participating site PI. Both cohorts, pts will be allowed to receive a 2nd treatment of 19-28z+ T cells if they benefited from the first infusion & did not experience any non-hematologic grade 4 toxicities.
  Interventions: Procedure: leukapheresis or collection of PBMCs; Drug: cyclophosphamide based chemotherapy regimens; Biological: modified T cells

INTERVENTIONS:
Procedure: leukapheresis or collection of PBMCs
Drug: cyclophosphamide based chemotherapy regimens
Biological: modified T cells

SUMMARY:
The purpose of this study is to test the safety of giving the patient special cells made from their own blood called "Modified T-cells". The goal is to find a safe dose of modified T-cells for patients whose leukemia has returned to the bone marrow.

DETAILED DESCRIPTION:
This is a phase I multicenter clinical trial for pediatric and young adult patients with relapsed/refractory CD19+ B-ALL. The T cell doses originally proposed in this study were based on doses administered safely in prior T cell adoptive therapy trials, but the dose has been modified based on the toxicities observed in adult patients with morphologic evidence of relapsed B-ALL treated on MSKCC IRB 09-114.

ELIGIBILITY:
Inclusion Criteria for Collection Arm of the protocol:

Age < 26 years, whose disease meets one of the following 3 criteria:

* VHR*
* Patients in 1st or subsequent marrow relapse (isolated or combined), at the time of relapse, during retrieval therapy, or after achievement of CR.
* Refractory disease *Definitions of VHR B-ALL include the following:

  * NCI HR-ALL and age ≥ 13 years at diagnosis
  * CNS-3 leukemia at diagnosis
  * Day 29/End of Induction BM MRD > 0.01%
  * Induction failure (M3 BM at Day 29/End of Induction)
  * Hypodiploidy (n< 44 chromosomes and/or a DNA index < 0.81)
  * t(9;22) ALL (Philadelphia Chromosome/Ph+ ALL)
  * t(17;19) ALL or Ph-Like ALL
  * MLL gene rearrangement
  * IKZF1 deletions
  * Intrachromosomal amplification of chromosome 21 (iAMP21) Please note patients that only meet the criteria for collection/storage of PBMCs will need to be reconsented prior to infusion of genetically modified T-cells.

Inclusion Criteria for Treatment Arm of this protocol:

* Patients must have a history of relapsed/refractory CD19+ B-ALL involving the marrow to be eligible for infusion of modified T cells.
* Please note ≥5% blasts by morphology, FISH/cytogenetics, molecular translocation and/or flow cytometry constitutes a bone marrow relapse on this protocol. Patients must also fulfill one of the following criteria to be eligible for infusion of modified T cells:

  * Second or greater (≥2) relapse
  * Early first marrow relapse (1st CR <18 months)
  * Intermediate/Late first marrow relapse (1st CR >18 months) with poor initial response (≥5% blasts by morphology and/or flow cytometry) following reinduction chemotherapy
  * Refractory Disease
  * Ineligible for HSCT as determined by the treating physician in consultation with the BMT service
  * Patient would not benefit from additional chemotherapy as determined by the treating physician
* KPS or Lansky score ≥ 60
* Pulmonary function (measured prior to conditioning chemotherapy):

  o > 90% oxygen saturation on room air by pulse oximetry.
* Renal Function (measured prior to conditioning chemotherapy):

  o Serum creatinine ≤2.0mg/dL for patients over 18 years or ≤2.5 x institutional ULN for age
* Hepatic Function (measured prior to conditioning chemotherapy):

  * AST ≤ 5 x the institutional ULN. Elevation secondary to leukemic involvement is not an exclusion criterion. Leukemic involvement will be determined by the presence of progressive relapse defined by escalating bone marrow or peripheral blood leukemia blasts within the previous month and the absence of initiation of know hepatotoxic medication (e.g. azoles).
  * Total bilirubin ≤ 2.5 x the institutional ULN

Exclusion Criteria for Collection of T cells/PBMCs:

* Karnofsky/Lansky performance status <60.
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation
* Patients with active HIV, hepatitis B or hepatitis C infection.
* Females who are pregnant

Exclusion Criteria for Treatment:

* Karnofsky/Lansky performance status <60.
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation
* Patients will be excluded if they have isolated extra-medullary relapse of ALL
* Females who are pregnant.
* Patients with active (grade 2-4) acute graft versus host disease (GVHD), chronic GVHD or an overt autoimmune disease (e.g. hemolytic anemia) following allo-HSCT requiring glucocorticosteroid treatment (>0.5 mg/kg/day prednisone or its equivalent) as treatment.
* Active central nervous system (CNS) leukemia, as defined by unequivocal morphologic evidence of lymphoblasts in the cerebrospinal fluid (CSF) within 7 days of treatment or symptomatic CNS leukemia (i.e. cranial nerve palsies or other significant neurologic dysfunction) within 28 days of treatment. Prophylactic intrathecal medication is not a reason for exclusion.

  o If the LP is traumatic (containing RBCs) and cannot be repeated the Steinherz/Bleyer ratio will be used to determined unequivocal evidence of CSF leukemia at the discretion of the treating physician.
* Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the treating investigator would pose an unacceptable risk to the subject.
* Prior neurologic toxicity to previous immunotherapy
* Preceding and/or ongoing organ dysfunction or other co-morbidity including but not limited to uncontrolled infection that would impair the patient's ability to endure known side effects of cytokine release syndrome or neurologic toxicity
* Recent prior therapy: Systemic chemotherapy less than 2 weeks prior to infusion or apheresis (6 weeks for clofarabine or nitrosoureas for apheresis) or radiation therapy less than or equal to 3 weeks prior to apheresis. Exceptions:

oThere is no time restriction in regard to prior intrathecal chemotherapy provided there is complete recovery from any acute toxic effects of such.

oSubjects receiving hydroxyurea or oral maintenance chemotherapy may be enrolled provided there has been no increase in dose for at least 2 weeks prior to starting apheresis or treatment.

oSubjects receiving steroid therapy at physiologic replacement doses only are allowed provided there has been no increase in dose for at least 2 weeks prior to starting apheresis or treatment.

oSubjects must have recovered from the acute side effects of their prior therapy, such that eligibility criteria are met. Cytopenias deemed to be disease-related and not therapy-related are exempt from this exclusion.

•Rapidly progressive disease that in the estimation of the treating physician would compromise ability to complete study therapy.

Max Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
safety | 1 year
  of gene-modified autologous T cells targeted to CD19 and infused into patients with relapsed/refractory B- ALL. Toxicities will be graded on a scale of 1 to 5 as described by the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. Adverse Events/Toxicities will be graded/attributed starting at time of T cell infusion and continue for up to 30 days or until modified T cells are no longer present.

SECONDARY OUTCOMES:
assess the persistence of modified T cells | 1 year
  Gene-modified T cells will be measured as per Table II from peripheral blood, bone marrow and/or lymph nodes. The percentage of gene-modified T cells T cells will be calculated and summarized at each follow-up time point. The data will be plotted over time to describe the time trend of T cell persistence.
the development of B cell aplasia | 1 year
  B cell aplasia will be measured as a surrogate marker for 19-28z+ T cell efficacy. Serum levels of normal B cells from peripheral blood and bone marrow aspirates will be monitored by FACS. The mean cell concentrations will be summarized and plotted against time.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Curran, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute:Dana- Farber/Children's Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Valtis YK, Lin C, Nemirovsky D, Devlin SM, Rejeski K, Curran KJ, Wang X, Shah NN, Jeyakumar N, Miller K, Zhang A, Kota VK, Al Darobi A, Muhsen IN, Sasine JP, Aldoss I, Advani AS, Reshef R, Chen EC, Kopmar NE, Tsai SB, Hilal T, Shah BD, Faramand RG, Solh MM, Tan V, Bezerra ED, Battiwalla M, Ramakrishnan A, Mathews J, Shaughnessy PJ, Mountjoy L, Hoeg RT, Dykes KC, Logan AC, Kumaran M, Schwartz MS, Tracy SI, Moore J, Odstrcil Bobillo S, Frey NV, Connor MP, Ladha A, Dholaria B, Sutherland KC, Roloff GW, Muffly LS, Park JH. CAR HEMATOTOX independently predicts outcomes after CD19 CAR-T therapy for acute lymphoblastic leukemia. Blood Adv. 2025 Oct 6:bloodadvances.2025017526. doi: 10.1182/bloodadvances.2025017526. Online ahead of print. PMID 41052404
- [Derived] Curran KJ, Margossian SP, Kernan NA, Silverman LB, Williams DA, Shukla N, Kobos R, Forlenza CJ, Steinherz P, Prockop S, Boulad F, Spitzer B, Cancio MI, Boelens JJ, Kung AL, Khakoo Y, Szenes V, Park JH, Sauter CS, Heller G, Wang X, Senechal B, O'Reilly RJ, Riviere I, Sadelain M, Brentjens RJ. Toxicity and response after CD19-specific CAR T-cell therapy in pediatric/young adult relapsed/refractory B-ALL. Blood. 2019 Dec 26;134(26):2361-2368. doi: 10.1182/blood.2019001641. PMID 31650176
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/